CLINICAL TRIAL: NCT05572580
Title: Evaluation of the German Version of a Validated Keratoconus Questionaire
Acronym: KORQ
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Opthalmology-008
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Keratoconus, Unspecified, Bilateral
MeSH Terms: conditions — Keratoconus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — the patients are asked to fill in a questionnaire

SUMMARY:
Keratoconus, which results in thinning of the cornea, affects mainly young patients. The causes are currently only partially known. The aim of this study is the evaluation of a keratoconus questionnaire in German. Until now this questionnaire is only in use in English.

Within the study patients will be asked to fill out a questionnaire. The questionnaire deals with issues that are influenced by keratoconus: Visual impairment and its impact on quality of life. This questionnaire (KORQ) is an already validated questionnaire in English. Within this study we would like to translate the questionnaire and validate it in German.

Within this study 50 patients will be included for the validation of the questionnaire. Based on previous studies evaluating the Keratoconus Questionnaire (KORQ) in other languages, a number of 50 patients has been shown to be sufficient for validation.

No control examination is necessary for this study.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus
* Signing of a written consent form for participation in the study

Exclusion Criteria:

* Difficulty in understanding patient information

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited in the keratoconus outpatient clinic as part of our routine checkups
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Validation of Keratoconus Outcome Research Questionnaire (KORQ) | at screening visit
  validation of a questionnaire in german language

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, Principal Investigator — Kepler University Hosiptal
Locations (1):
- Kepler University Klinik, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided